CLINICAL TRIAL: NCT01599884
Title: Effects of High-Dose N-Acetylcysteine on Respiratory Health Status in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Bronchitis: A Randomized, Placebo-Controlled Trial-1
Brief Title: N-Acetylcysteine for Patients With COPD and ChronicBronchitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Veterans Research and Education (Other)
Responsible Party: Principal Investigator, Dennis Niewoehner, Staff physician, Center for Veterans Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MVMREF-001; NCT01639963 (obsolete NCT alias)
Record Dates: First submitted 2012-05-15; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: Chronic obstructive pulmonary disease; Chronic bronchitis; N-acetylcysteine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Active Comparator): N-acetylcysteine, 1800 mg twice daily
  Interventions: Drug: N-acetylcysteine
- Sugar pill (Placebo Comparator): Identical to active drug
  Interventions: Drug: Oral acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 1800 mg twice daily for 8 weeks
  Arms: N-acetylcysteine
Drug: Oral acetylcysteine — Identical placebo pills twice daily for 8 weeks
  Arms: Sugar pill

SUMMARY:
N-acetylcysteine (NAC) is described as having mucolytic and antioxidant properties. It is widely prescribed for patients with chronic obstructive pulmonary disease (COPD), particularly for those who have accompanying symptoms of chronic cough and sputum production. Randomized, placebo controlled indicate that it is safe and that it may have some clinical benefit when used at relatively low doses. It is postulated that substantially higher doses of NAC will be well-tolerated and will provide better symptom control while also decreasing blood makers of oxidant stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Capability to provide written informed consent
  * Age ≥ 40 years and ≤ 85 years
  * FEV1/FVC ratio (post bronchodilator) < 70%
  * FEV1 (post bronchodilator) < 65%
  * Presence of chronic cough and sputum production defined as the following:
* Presence of chronic cough and sputum will be defined by responses to the first two questions on the SGRQ (see Appendix A). Subjects who respond positively to both question 1 (cough) and question 2 (sputum) on the SGRQ as either "several days per week" or "almost every day" will be eligible

  * Current or former smoker with lifetime cigarette consumption of at least 10 pack-years
  * Negative serum pregnancy test at the baseline visit if patient is a pre-menopausal female (menopause defined as absence of a menstrual cycle in the last 12 months)
  * Must be fluent in speaking the English language
* Exclusion Criteria

  * Not fully recovered for at least 30 days from a COPD exacerbation characterized by typical symptoms and treated with antibiotics or prednisone
  * Known allergy or sensitivity to NAC or albuterol
  * Any patient with unstable cardiac disease
  * Any patient with a documented history of uncompensated congestive heart failure in the last 2 years
  * Clinical diagnosis of asthma, bronchiectasis, cystic fibrosis, or severe alpha-1 antitrypsin deficiency
  * Active lung cancer or history of lung cancer if it has been less than 2 years since lung resection or other treatment. If history of lung cancer, must have no evidence of recurrence in the 2 years preceding the baseline visit.
  * Undergoing active treatment for malignancy except for hormonal therapy (i.e. prostate cancer, breast cancer) or non-metastatic skin cancer and are not symptomatic
  * Chronic kidney disease with an estimated GFR of < 30 ml/min. GFR will be estimated using the Modification of Diet in Renal Disease (MDRD) formula
  * History of cirrhosis with evidence of portal hypertension (ascites, chronic edema)
  * Participation in a pulmonary rehabilitation program or completion within past 6 weeks
  * Prisoners or institutionalized patients
  * Participation in another study involving an investigational product within 30 days of the baseline visit
  * Pregnant or breast-feeding patients.
  * Use of guaifenesin in the last 30 days
  * Currently on long acting nitrates for angina or heart failure
  * Abnormalities in screening blood work defined as:
* WBC < 3.0 or > 15.0 K/cmm
* Hemoglobin < 9.0 or > 17.0 gm/dl
* Platelets < 75 or > 400 K/cmm
* ALT > 3 times the upper limit of normal
* INR > 1.5 unless on warfarin therapy o Any concomitant condition that might endanger the patient through participation in the study or interfere with study procedures, as assessed by the investigator

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the St. George's Respiratory Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Niewoehner, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States